CLINICAL TRIAL: NCT06726980
Title: Effects of Dextrose Versus Saline Infusion on Intrathecal Morphine-Induced Postoperative Nausea and Vomiting During Gynecological Abdominal Surgeries: Randomized Controlled Double-blind Study
Status: Not yet recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Fareed Fathy Wadea, resident doctor at Anaesthesia, Intensive Care and Pain Management Faculty of Medicine, Assiut University, Assiut University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: Dextrose vs Saline Gyn surg
Record Dates: First submitted 2024-12-05; First posted 2024-12-10 (Actual); Last update posted 2024-12-10 (Actual); Status verified 2024-12

CONDITIONS: Gynecological Abdominal Surgeries
Keywords: Nausea; Vomiting; Dextrose
MeSH Terms: conditions — Nausea; Vomiting | interventions — Saline Solution

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (3):
- group I (Placebo Comparator): patients will receive infused IV 0.9 % saline
  Interventions: Drug: 0.9% saline
- Study group II (Experimental): patients will receive 5 % dextrose infusion
  Interventions: Drug: dextrose 5%
- Study group III (Experimental): patients will receive 10 % dextrose infusion (25gm/ 250 mL)
  Interventions: Drug: Dextrose 10%

INTERVENTIONS:
Drug: dextrose 5% — patients will receive 5 % dextrose infusion
  Arms: Study group II
Drug: Dextrose 10% — patients will receive 10 % dextrose infusion (25gm/ 250 mL)
  Arms: Study group III
Drug: 0.9% saline — patients will receive infused IV 0.9 % saline
  Arms: group I

SUMMARY:
Neuraxial anesthesia, which includes epidural anesthesia and intrathecal anesthesia, is a frequent anesthetic approach for cesarean delivery and other lower abdominal and lower limb anesthetic procedures.

Neuraxial morphine (intrathecal or epidural administration) provides high-quality analgesia after gynecological abdominal surgeries.

the aim of the study is to compare the effects of intraoperative infusion of dextrose 5 % and 10 % versus normal saline 0.9 % on the incidence of intrathecal morphine-induced postoperative nausea and vomiting (PONV) in women undergoing gynecological abdominal surgeries. (Neuraxial anesthesia).

DETAILED DESCRIPTION:
The use of intrathecal opioids for postoperative analgesia was introduced in 1979. There have been many pharmacodynamic and pharmacokinetic studies of intrathecal opioids and the mechanism of action-producing analgesic effects by direct action at the spinal cord level. The addition of intrathecal opioids to bupivacaine for spinal anesthesia may provide clinical advantages such as improved intraoperative conditions and postoperative analgesia. Adverse effects range from nausea and vomiting that, although not life-threatening, are major nuisances to the patient, to more severe effects, including sedation and life-threatening respiratory depression.

Nausea is an unpleasant sensation causing discomfort in the stomach area which gives the feeling of the impending need to vomit or retch. It is often a transient sensation which is frequently followed by active retching or tachycardia and increased salivation. Vomiting is the involuntary, forceful expulsion of the contents of the stomach through the mouth and/or nose. The incidence of these side effects varies from 30-80 % after elective surgery depending on the type of anesthesia and surgery as well as predisposing patient risk factors.

Postoperative nausea and vomiting (PONV) describes nausea and/or vomiting or retching occurring in the post-anesthesia care unit (PACU) or during the first 24-48 hours after surgery. Post-discharge nausea and vomiting (PDNV) refers to symptoms that occur after discharge from the hospital or surgical care facility. Not only is PONV a distressing complication from the patient's perspective but also it can result in dehydration, electrolyte imbalance, acid base imbalance, pulmonary aspiration, pneumothorax, hypoxia, esophageal rupture, increased intracranial pressure, suture rupture, wound dehiscence, bleeding, delay in the ability to resume oral intake, prolonged PACU and/or hospital stay, fatigue, anxiety, unanticipated hospital admission or readmission, and increased medical costs. The distressing symptoms of PONV/PDNV also contribute to patient dissatisfaction with their surgical experience. PONV prophylaxis is economically beneficial for the hospital when a rational multimodal program is implemented based on patient and procedural risk factors.

Enhanced recovery programs in surgical patients and the promotion of day case surgery both require and include adequate prophylaxis of PONV. There are dozens of different anti-emetic drugs, mostly within the drug classes of 5- hydroxytryptamine-3 (5HT3), dopamine-2 (D2) and neurokinin-1 (NK1) receptor antagonists, corticosteroids, antihistamines and anticholinergics. Varying adverse effects have been attributed to the six different substance classes, such as headache and constipation (5-HT3 receptor antagonists); extrapyramidal symptoms, sedation, arrhythmia and QT prolongation (D2 receptor antagonists); hyperglycemia, immunosuppression and poor wound healing (corticosteroids); drowsiness, dry mouth and urinary difficulties (antihistamines); and dry mouth and visual disturbances (anticholinergics).

In addition to pharmacological therapy, recent studies are assessing the impact of fluid therapy in the prevention of PONV, finding that the use of crystalloids in ASA I and II patients receiving general anesthesia reduces the risk of postoperative nausea. and a preventive effect of vomiting during the first 24 hrs post-surgery[15]. Another fluid therapy strategy for PONV is the administration of colloids, which has had a superior effect in preventing PONV than the administration of crystalloids in patients undergoing lower abdominal surgery who received general anesthesia for 3 hours or more[16]; however, these results are not the same in patients who received general anesthesia for less than 3 hours. On the other hand, the administration of bolus glucose solution is still very controversial, since some results show that it does not reduce PONV [17], while Chisaki et al. (2020) reported its usefulness in reducing postoperative nausea, but not vomiting.

These last fluid therapy recommendations should be handled with caution, since the risk of serious adverse events resulting from the supplementary administration of intravenous crystalloids and colloids is unknown, and it is not clear whether patients are at risk of being readmitted to the hospital postoperatively due to these interventional measures.

ELIGIBILITY:
Inclusion Criteria:

* Age: 20 - 60 years. Females of American Society of Anesthesiologists (ASA) class I or II physical status.

Elective gynecological abdominal surgeries under intrathecal anesthesia.

Exclusion Criteria:

* Patient refusal. Patients with a history of PONV, smoking, motion sickness or diabetes mellitus. Significant organ dysfunctions (e.g., cardiac, respiratory, renal, or liver disorders).

Morbid obesity (BMI >35 kg/m²). Patients with known hypersensitivity to morphine or amide local anesthetics. Patients with any contraindication for intrathecal anesthesia, e.g. coagulopathy.

Emergency operations. Psychiatric disorders or patients who are unable to understand the verbal rating scale.

Failed or unsatisfactory intrathecal block. Patients currently receiving opioids, steroids, antiemetic drugs or chemotherapy, pregnant females, and those with abnormal blood glucose on the morning of surgery.

Ages: 20 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes — female
Enrollment: 63 (Estimated)
Dates: Start 2025-01-01 (Estimated); Primary Completion 2026-01-01 (Estimated); Study Completion 2026-02-01 (Estimated)

PRIMARY OUTCOMES:
Incidence of postoperative nausea and vomiting( PONV) | 24 hours
  Incidence of PONV during the first postoperative 24 hours

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Yokoyama C, Mihara T, Kashiwagi S, Koga M, Goto T. Effects of intravenous dextrose on preventing postoperative nausea and vomiting: A systematic review and meta-analysis with trial sequential analysis. PLoS One. 2020 Apr 20;15(4):e0231958. doi: 10.1371/journal.pone.0231958. eCollection 2020. PMID 32310996
- [Background] Kim HJ, Choi SH, Eum D, Kim SH. Is perioperative colloid infusion more effective than crystalloid in preventing postoperative nausea and vomiting?: A systematic review and meta-analysis. Medicine (Baltimore). 2019 Feb;98(7):e14339. doi: 10.1097/MD.0000000000014339. PMID 30762734
- [Background] Jewer JK, Wong MJ, Bird SJ, Habib AS, Parker R, George RB. Supplemental peri-operative intravenous crystalloids for postoperative nausea and vomiting: an abridged Cochrane systematic review. Anaesthesia. 2020 Feb;75(2):254-265. doi: 10.1111/anae.14857. Epub 2019 Sep 19. PMID 31536172
- [Background] Wiesmann T, Kranke P, Eberhart L. Postoperative nausea and vomiting - a narrative review of pathophysiology, pharmacotherapy and clinical management strategies. Expert Opin Pharmacother. 2015 May;16(7):1069-77. doi: 10.1517/14656566.2015.1033398. Epub 2015 Apr 12. PMID 25866213
- [Background] Metz A, Hebbard G. Nausea and vomiting in adults--a diagnostic approach. Aust Fam Physician. 2007 Sep;36(9):688-92. PMID 17885699
- [Background] Balaban CD, Yates BJ. What is nausea? A historical analysis of changing views. Auton Neurosci. 2017 Jan;202:5-17. doi: 10.1016/j.autneu.2016.07.003. Epub 2016 Jul 16. PMID 27450627
- [Background] Koju RB, Gurung BS, Dongol Y. Prophylactic administration of ondansetron in prevention of intrathecal morphine-induced pruritus and post-operative nausea and vomiting in patients undergoing caesarean section. BMC Anesthesiol. 2015 Feb 17;15:18. doi: 10.1186/1471-2253-15-18. PMID 25971957